CLINICAL TRIAL: NCT05950711
Title: Ketamine-Assisted Mindfulness-Based Cognitive Therapy for Depression: A Pilot Study
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Ohio State University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020H0374
Record Dates: First submitted 2023-04-03; First posted 2023-07-18 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Major Depressive Disorder
Keywords: Ketamine; Mindfulness-Based Cognitive Therapy; Major depressive disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Ketamine

STUDY DESIGN:
Intervention Model Description: Open Label Feasibility Study of an Intervention Without a Control Group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Ketamine-MBCT Intervention (Experimental): One Arm: Combination of MBCT with a single ketamine infusion
  Interventions: Other: Combination use of MBCT and IV Ketamine

INTERVENTIONS:
Other: Combination use of MBCT and IV Ketamine — Group with Major Depression who will receive a single dose of IV Ketamine embedded within a course of MBCT.

SUMMARY:
The purpose of this study is to assess the feasibility of combining IV ketamine, a rapid acting antidepressant, with a course of Mindfulness-Based Cognitive Therapy (MBCT), for the initial and maintenance treatment of depression.

DETAILED DESCRIPTION:
The purpose of this study is to assess the feasibility of combining IV ketamine, a rapid acting antidepressant, with a course of Mindfulness-Based Cognitive Therapy (MBCT), for the initial and maintenance treatment of depression. Both ketamine and MBCT are used for treatment of depression, however, the combination of ketamine and psychotherapy has been studied mostly for drug addiction. Despite its rapid onset and effectiveness for depression, ketamine is most effective in the short term. MBCT is a therapeutic approach that combines cognitive behavioral techniques (CBT) with mindfulness strategies in order to help individuals better understand and manage their thoughts and emotions that can both decrease and prevent the relapse of the symptoms of depression. The aim of this pilot study is to embed one infusion of ketamine in the MBCT treatment. Our hypothesis is that the initial positive effect of ketamine will help patients engage in the behavioral therapy, which itself provides cognitive/emotion control tools to prevent relapses of depression.

ELIGIBILITY:
Inclusion Criteria:

* Adults age 18-65
* A current diagnosis of major depressive disorder according to DSM-5 criteria per MINI interview
* Moderate to severe level of current depressive symptoms (MADRS score ≥20)
* Failure of at least one adequate trial of antidepressant medication (defined as: therapeutic doses of antidepressant medication for ≥ 6 weeks)
* No adverse reactions to ketamine
* Capacity to consent and comply with study procedures, including sufficient proficiency in English

Exclusion Criteria:

* Meets DSM-5 criteria for bipolar disorder, schizophrenia, any psychotic illness, including substance-induced psychosis, active PTSD, dissociative disorders and current substance-induced mood disorder, OCD, eating disorder, panic disorder.
* Suicide attempt in the past 4 weeks or current risk of suicide
* Current alcohol or drug substance use disorder according to DSM-5
* Cognitive- or intellectual impairments which would interfere with participation in MBCT or assessments including meeting criteria for Delirium, Dementia, Amnesia, Cognitive Disorders,
* Personality Disorders (borderline, antisocial, paranoid, schizoid, histrionic) that may interfere with treatment
* Previous participation in MBCT or MBSR group
* Pregnant or planning to become pregnant during the study period
* Heart disease as indicated by history, abnormal ECG, previous cardiac surgery.
* Hypertension (>160/100)
* Unstable physical disorders which might make participation hazardous such as history of AIDS, known lab abnormalities, active hepatitis or other liver disease with elevated transaminase levels (< 2-3 X upper limit of normal will be considered acceptable if PT/PTT is normal), renal failure (creatinine > 2, BUN >40), or untreated diabetes.
* Previous history of ketamine misuse or abuse, or a history of an adverse reaction/experience with prior exposure to ketamine
* BMI > 32
* History of documented obstructive sleep apnea
* On psychotropic or other medications whose effect could be disrupted by participation in the study or not allowed during the study (such as monoamine oxidase inhibitors).
* Patient unable or unlikely to comply with the study protocol or for any other conditions that might indicate that the patient is unsuitable for the study as judged by the investigator
* Positive urine drug screen, except for marijuana or benzodiazepine if prescribed.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2022-03-30 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Change in MADRS score | 12 months
  Response defined a ≥50% reduction in depressive symptoms as measured of standardized measures; remission defined as decrease of depression scores below cut-off for the scale

SECONDARY OUTCOMES:
Change in PHQ9 score | 12 months
  Response defined a ≥50% reduction in depressive symptoms on the PHQ9
Correlation between MADRS/PHQ9 score and Mystic experience scores | 12 months
  analysis of possible correlation between depression scales scores and mystic experience during the ketamine infusion

CONTACTS AND LOCATIONS:
Locations (1):
- Harding Hospital, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share our data with other researchers